CLINICAL TRIAL: NCT03131076
Title: Intraduktaalisen Papillaarisen Musinoosisen Neoplasian Vuoksi Seurannassa Olevien Potilaiden elämänlaatu
Brief Title: Quality of Life Assessment in Patients Who Are Under Surveillance for IPMN
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Heini Nieminen, licensed physician, Helsinki University Central Hospital
Other Study IDs: IPMN Quality of life
Record Dates: First submitted 2017-04-07; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: IPMN; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: IPMN follow up — Follow up with MRI and laboratory blood tests

SUMMARY:
Over 500 patients were participating in the IPMN follow up between september 2014 and august 2016 at the Helsinki University Hospital. In this study we are going to determine the effects of the IPMN surveillance on the quality of life and anxiety levels of the patients.

DETAILED DESCRIPTION:
Intraductal papillary mucinous neoplasm (IPMN) is a cystic neoplasm of the pancreas. The incidence of the tumors has increased during the last years. Some of the IPMN-tumors develop over time increasing dysplasia and at the end IPMN associated carcinoma. All IPMN-patients are kept under surveillance because of the cancer risk. This follow up can last decades and includes MRI and blood samples every 6 to 12 months. This is very expensive and the effects on the patients quality of life have not been studied before to our knowledge.

This study determines the effects of the surveillance on the patients quality of life and anxiety levels. The study will be conducted by 15D- quality of life -questionnaire and state-trait anxiety inventory (STAI) -questionaire. Both will be send to the patients before a IPMN follow up MRI and 3 months later. It is anticipated that the anxiety and the effect on the quality of life would be the highest right before the MRI and would normalize a few months after the MRI.

ELIGIBILITY:
Inclusion Criteria:

* all patients under IPMN surveillance

Exclusion Criteria:

* no exclusion criteria, all patients under IPMN surveillance are included

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients under IPMN follow up
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the quality of life and anxiety | Before and 3 months after IPMN follow up MRI
  15D quality of life and STAI -questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Heini Nieminen, Principal Investigator — Helsinki Universtity Hospital

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.

REFERENCES:
- [Derived] Nieminen H, Roine R, Ristimaki A, Lantto E, Valimaa N, Kirveskari E, Sintonen H, Haglund C, Seppanen H. Health-related quality of life and anxiety levels among patients under surveillance for intraductal papillary mucinous neoplasm. BMC Gastroenterol. 2023 Jan 16;23(1):14. doi: 10.1186/s12876-023-02639-0. PMID 36647007